CLINICAL TRIAL: NCT01413256
Title: Allergenic Effect of Ambrosia in Israel
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: EDUARDO SHAHAR, RAMBAM MEDICAL CENTER
Other Study IDs: 0015-11-RMB
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-08

CONDITIONS: Allergy; Ambrosia; Ragweed
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
Background:

Respiratory allergic reaction causes great suffering to millions of people worldwide. One of the most known allergen- is the pollen from vegetation, ragweed. Genus Ambrosia Ambrosia belonged to the complex ragweed flowers are pollinated by the wind and the plant's male flowers produce large quantities of small grains of pollen and airborne over long distances and those causes allergic reactions. The plant blooms between June and October, creating a second wave after wave of allergy caused by spring blossoms.

This plant originated in North America has invaded many areas in Europe and in recent years, taking over large areas in Israel, Hula Valley and northern Acre Emek Hefer for a pen and layers to the south. After ragweed plants are based in particular they spread quickly and invade agricultural fields and significantly reduce the crop.

High allergenic ragweed is a health hazard to humans. Ragweed plant investigated many aspects of North America and Europe in recent decades and extensive literature on ambrosia, but this is the first time ragweed study focuses on Israel.

Working hypothesis and aims:

Goal of this study is to identify the existence and nature of the sensitivity distribution of ragweed in Israel.

Importance of research:

A. Ragweed allergen testing and comparing the effect of exposure to plants on the sensitivity of the allergic Israeli patients

B. The inclusion of ragweed allergen in the diagnostic and therapeutic panel

ELIGIBILITY:
Inclusion Criteria:

* respiratory allergic patients

Exclusion Criteria:

* non respiratory allergic patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: respiratory allergic patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)